CLINICAL TRIAL: NCT03006874
Title: A Double Blind, Randomized, Active-controlled, Phase 3 Study to Confirm the Safety and Efficacy of CJ-12420 in Patients With Erosive Esophagitis
Brief Title: Study to Confirm the Safety and Efficacy of CJ-12420 in Patients With Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_APA_304
Record Dates: First submitted 2016-06-14; First posted 2016-12-30 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — tegoprazan; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CJ-12420 50mg QD (Experimental): CJ-12420 50mg tablet, once daily, oral administration for up to 8 weeks.
  Interventions: Drug: CJ-12420 50mg QD
- CJ-12420 100mg QD (Experimental): CJ-12420 100mg tablet, once daily, oral administration for up to 8 weeks.
  Interventions: Drug: CJ-12420 100mg QD
- Esomeprazole 40mg (Active Comparator): Esomeprazole 40mg, tablet. once daily, oral administration for up to 8 weeks.
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: CJ-12420 100mg QD — CJ-12420 100mg tablets will be orally administered, once daily, for up to 8 weeks. For subjects whose erosive esophagitis is not endoscopically healed at Week 4, subjects will receive additional 4 week treatment of CJ-12420 100mg.
  Other Names: Tegoprazan Tab.
  Arms: CJ-12420 100mg QD
Drug: Esomeprazole 40mg — Esomeprazole 40mg tablets will be orally administered, once daily, for up to 8 weeks. For subjects whose erosive esophagitis is not endoscopically healed at Week 4, subjects will receive additional 4 week treatment of Esomeprazole 40mg.
  Other Names: Nexium Tab.
  Arms: Esomeprazole 40mg
Drug: CJ-12420 50mg QD — CJ-12420 50mg tablets will be orally administered, once daily, for up to 8 weeks. For subjects whose erosive esophagitis is not endoscopically healed at Week 4, subjects will receive additional 4 week treatment of CJ-12420 50mg.
  Other Names: Tegoprazan Tab.
  Arms: CJ-12420 50mg QD

SUMMARY:
The purpose of this study is to confirm the efficacy of CJ-12420, Once daily (QD), compared to esomeprazole in patients with erosive esophagitis classified as Los Angeles (LA) classification grades A to D at Week 8.

DETAILED DESCRIPTION:
This is a double blind, randomized, active controlled, phase 3 study. Subjects will be randomly assigned to one of the three treatment groups (CJ-12420 50mg, CJ-12420 100mg, esomeprazole 40mg).

All subjects will be asked to take three tablets at the same time each day throughout the study, and also all subjects will be asked to record daytime and nighttime symptom in a subject diary on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 20 and 75 years
2. Endoscopically confirmed erosive esophagitis as defined by LA Classification Grading System (A-D) within 14 days prior to randomization
3. Subjects who had experienced heartburn and regurgitation within 7 days before visit 1
4. Subjects who is able to understand and follow the instructions and is willing to participate throughout the entire study
5. Subjects who voluntarily signed written informed consent form
6. Subjects who agreed to use medically acceptable contraceptives during the period of study

Exclusion Criteria:

1. Subjects who cannot undergo EGD
2. Subjects who have esophageal stenosis, ulcer stenosis, gastroesophageal varices, Barrett's esophagus, active gastric ulcer, gastrointestinal bleeding or malignant tumor confirmed by EGD
3. Subjects who have warning symptoms of malignant gastrointestinal tract such as odynophagia, severe dysphagia, bleeding, weight loss, anemia, or bloody stool
4. Subjects with eosinophilic esophagitis
5. Subjects diagnosed with primary esophageal motility disorder, IBS, IBD, etc. or with suspected IBS in the last 3 months
6. Subjects who have a history of gastric acid suppression surgery or upper gastrointestinal, esophageal surgery
7. Subjects who have AIDS or Hepatitis
8. Subjects who take antipsychotic drugs, antidepressant drug, antianxiety drug
9. Subjects who take gastric acid suppression like PPI within 2 weeks to EGD
10. Subjects who take medications related to reflux esophagitis more than 2 times within 1 weeks to EGD
11. Requirement of persistent daily use of drugs that may cause an ulcer such as nonsteroidal anti-inflammatory drugs(NSAIDs) or aspirin during the course of the study
12. Pregnant or lactating women
13. Subjects with the following clinically significant laboratory abnormalities
14. Subjects with the following clinically significant ECG abnormalities
15. Sollinger-Ellison syndrome patients
16. Subjects with a history of malignant tumor
17. Subjects with a history of clinically significant hepatic, renal, cardiovascular, respiratory, endocrine and CNS system disorder
18. Subjects with a history of hypersensitivity to the active ingredient or excipients of the study drug, etc
19. Scheduled surgery requiring hospitalization or requirement of surgical treatment during study participation
20. Subjects who participated in the other clinical trial within 4 weeks prior to randomization
21. Subjects who are judged unsuitable to participate in the study in the opinion of the investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Cumulative healing rate of erosive esophagitis at 8-week | 8 week

SECONDARY OUTCOMES:
Healing rate of erosive esophagitis at 4-week | 4-week
Symptom assessment by subject diary | 4-week or 8-week
Symptom assessment by questionnaire | 4-week or 8-week

CONTACTS AND LOCATIONS:
Overall Officials: Poong Ryul Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No